CLINICAL TRIAL: NCT04495296
Title: A Phase I/IIa Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of TST001 - Claudin18.2 Monoclonal Antibody in the Treatment of Locally Advanced or Metastatic Solid Tumors
Brief Title: A Trial to Evaluate Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of TST001 in Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Transcenta Therapeutics Co., Ltd. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TST001-1002
Record Dates: First submitted 2020-07-23; First posted 2020-07-31 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Oxaliplatin; Capecitabine; Paclitaxel; Gemcitabine; Cisplatin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- dose escalation Q2W (Experimental): Dosed every 2 weeks IV with TST001, multiple dose levels will be tested.
  Interventions: Drug: TST001
- dose escalation Q3W (Experimental): Dosed every 3 weeks IV with TST001, multiple dose levels will be tested.
  Interventions: Drug: TST001
- Cohort A (Experimental): Participants with gastric or gastroesophageal junction cancers and CLDN18.2 expression
  Interventions: Drug: TST001
- Cohort B (Experimental): Participants with ductal adenocarcinoma of pancreas and CLDN18.2 expression and CLDN18.2 expression
  Interventions: Drug: TST001
- Cohort E (Experimental): Participants with advanced or metastatic solid tumors other than G/GEJ adenocarcinoma and CLDN18.2 expression
  Interventions: Drug: TST001
- Cohort C (Experimental): Participants with HER2 negative or unknown locally advanced or metastatic G/GEJ adenocarcinoma
  Interventions: Drug: TST001; Drug: Oxaliplatin; Drug: Capecitabine
- Cohort D (Experimental): Participants with locally advanced or metastatic G/GEJ adenocarcinoma
  Interventions: Drug: TST001; Drug: Paclitaxel
- Cohort F (Experimental): Participants with locally advanced or metastatic biliary tract cancer
  Interventions: Drug: TST001; Drug: Gemcitabine; Drug: Cisplatin
- Cohort G (Experimental): Participants with HER2 negative or unknown locally advanced or metastatic G/GEJ adenocarcinoma
  Interventions: Drug: TST001; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Nivolumab
- Cohort H (TST001 plus nivolumab) (Experimental): Participants with locally advanced or metastatic G/GEJ adenocarcinoma
  Interventions: Drug: TST001; Drug: Nivolumab

INTERVENTIONS:
Drug: TST001 — TST001 will be administered by specified doses on specified day
Drug: Oxaliplatin — Oxaliplatin will be administered by specified doses on specified day
  Arms: Cohort C; Cohort G
Drug: Capecitabine — Capecitabine will be administered by specified doses on specified day
  Arms: Cohort C; Cohort G
Drug: Paclitaxel — Paclitaxel will be administered by specified doses on specified day
  Arms: Cohort D
Drug: Gemcitabine — Gemcitabine will be administered by specified doses on specified day
  Arms: Cohort F
Drug: Cisplatin — Cisplatin will be administered by specified doses on specified days Oxaliplatin will be administered by specified doses on specified day Drug: Capecitabine Capecitabine will be administered by specified doses on specified day
  Arms: Cohort F
Drug: Nivolumab — Nivolumab will be administered by specified doses on specified day
  Arms: Cohort G; Cohort H (TST001 plus nivolumab)

SUMMARY:
This is an open-label, multi-center, Phase I trial of TST001. Subjects with locally advanced or metastatic solid tumors will be enrolled. The study will consist of two parts: Part A is dose escalation and dose expansion phase for mono-therapy, and Part B is dose escalation and dose expansion phase for combination therapy in gastric, gastroesophageal junction(G/GEJ) and biliary tract cancer, etc.

DETAILED DESCRIPTION:
There are two parts in the study. Part I is mono-therapy dose escalation and dose expansion study, and Part II is dose escalation and dose expansion study of combination therapy.

The dose escalation study will be conducted utilizing 3+3 design with two dosing regimens, i.e. "once every 2 weeks (Q2W)" and "once every 3 weeks (Q3W)".

After MTD/RP2D determined, three cohorts may be included in the expansion plan, with about 30 (20-40) subjects with positive CLDN18.2 expression be treated in each cohort, as shown below (during the study, the treatment cohorts may be adjusted or added based on the clinical and pre-clinical study data).

Approximately 320-540 treated subjects in total

ELIGIBILITY:
Inclusion Criteria:

The subjects who meet all inclusion criteria can be enrolled into the trial:

1. Sign the Informed Consent Form (ICF) voluntarily, understand the study and be willing and able to comply with all study procedures;
2. Male or female ≥ 18 years at signing the ICF;
3. Suffer from histologically confirmed locally unresectable advanced or metastatic solid tumors and meet the criteria of corresponding cohort as follows:

   Part I - Mono-therapy dose escalation and expansion phase:
   1. Mono-therapy dose escalation study: The subjects who have no option of or are intolerable to SOC.
   2. Mono-therapy dose expansion study: The subjects with positive CDLN18.2 expression in tumor tissue (defined as CLDN18.2 membranous staining ≥1+ in ≥10% of tumor cells by immunohistochemistry (IHC) in the central laboratory) confirmed by the central laboratory at enrollment. The dose expansion study may include the following 3 cohorts:

   Cohort A: Subjects with G/GEJ adenocarcinoma who have no option of or are intolerable to SOC; Cohort B: Subjects with ductal adenocarcinoma of pancreas who have no option of or are intolerable to SOC; Cohort E: Subjects with other locally advanced or metastatic solid tumors excluding G/GEJ adenocarcinoma (limited to biliary tract neoplasms, lung adenocarcinoma or colorectal cancer) who have no option of or are intolerable to SOC; Part II - Dose escalation and expansion phase for combination medication
   1. Dose escalation study of combination medication (dose escalation part):

      Cohort C/G: Subjects with HER2 negative or unknown G/GEJ adenocarcinoma who have not received prior systemic chemotherapy. The subjects who have completed neoadjuvant or adjuvant chemotherapy within at least 6 months prior to the initial dosing of the study can be enrolled.

      Cohort D: The subjects with G/GEJ adenocarcinoma who have received at least prior first-line systemic chemotherapy; Cohort F: The subjects with biliary neoplasm who have not received prior systematic chemotherapy. The subjects who have completed neoadjuvant or adjuvant chemotherapy within at least 6 months prior to the initial dosing of the study can be enrolled.

      Cohort H: The subjects with G/GEJ adenocarcinoma who have received at least prior second-line systemic chemotherapy;
   2. Dose expansion study of combination medication (dose expansion part):

   The subjects with positive CDLN18.2 expression in tumor tissue confirmed by the central laboratory will be enrolled as follows:

   Cohort C/G: Subjects with HER2 negative or unknown G/GEJ adenocarcinoma who have not received prior systemic chemotherapy. The subjects who have completed neoadjuvant or adjuvant chemotherapy within at least 6 months prior to the initial dosing of the study can be enrolled.

   Cohort D: The subjects with G/GEJ adenocarcinoma who have received at least prior first-line systemic chemotherapy; Cohort F: The subjects with biliary neoplasm who have not received prior systematic chemotherapy. The subjects who have completed neoadjuvant or adjuvant chemotherapy within at least 6 months prior to the initial dosing of the study can be enrolled.

   Cohort H: The subjects with G/GEJ adenocarcinoma who have received at least prior second-line systemic chemotherapy;
4. ECOG performance status of 0-1;
5. Life expectancy ≥ 3 months;
6. The results of laboratory examinations at screening must meet all the following criteria:

   1. Absolute neutrophil count (ANC) ≥ 1.5×109/L;
   2. Absolute white blood cell (WBC) count ≥2.5×109/L;
   3. Platelets ≥ 100×109/L;
   4. Haemoglobin ≥ 9 g/dL;
   5. International normalized ratio (INR) ≤ 1.5 times upper limit of normal (ULN) / or activated partial thromboplastin time (APTT) ≤ 1.5 times ULN (for the test without anticoagulant);
   6. INR ≤ 2.5 times ULN / or APTT ≤ 2.5 times ULN (for the test with anticoagulant);
   7. Total bilirubin <= 1.5 x ULN (except participants with Gilbert Syndrome who must have a total bilirubin level of < 3.0 mg/dL).;
   8. AST and ALT ≤ 2.5 times ULN (≤ 5 times ULN for subjects with hepatic cancer or liver metastases); ALT/AST ≤ 3xULN regardless of liver metastasis for cohort G and H only;
   9. Albumin ≥ 30g/L;
   10. Serum creatinine ≤ 1.5 times ULN, or creatinine clearance rate ≥ 60 ml/min (creatinine clearance rate will be calculated using Cock-croft-Gault Equation);
7. Male and female of childbearing age should agree to take effective contraception measures (refer to Appendix 3. Contraception) from signing the ICF till at least 120 days post the last dose of TST001 and other study drugs except nivolumab; female of childbearing age should agree to take effective contraception measures (refer to Appendix 3. Contraception) from signing the ICF till at least 5 months post the last dose of nivolumab; Serum β-HCG test for women of childbearing age within 72 hours prior to the initial dosing must be negative;
8. (For dose expansion phase only) At least one measurable lesion conforming to per RECIST v1.1;

Exclusion Criteria:

The subjects who meet any one of the following criteria will be excluded from participation in this study:

1. The subjects with locally advanced or metastatic G/GEJ adenocarcinoma who are supposed to be enrolled into the combination therapy cohorts with CAPOX and CAPOX+nivolumab (Cohort C and G) have previously received systemic chemotherapy; and the subjects in the Cohort G have previously received PD1/PD-L1/CTLA4 antibody treatment. The subjects will be eligible provided that they have completed neoadjuvant or adjuvant chemotherapy at least 6 months prior to the initial dosing of the study; The subjects with locally advanced or metastatic G/GEJ adenocarcinoma who are supposed to be enrolled into the combination therapy cohort with paclitaxel (Cohort D) have previously received taxane drugs.
2. The subjects who previously received radiotherapy within 4 weeks prior to the initial dosing of the investigational drug (the subjects who previously received local radiotherapy for bone metastases treatment within 4 weeks with the radiotherapy related AE resolved to ≤ Grade 1 will be eligible);
3. The subjects who previously received other systematic anti-tumor drug therapies within 4 weeks or 5 half-lives prior to the initial dosing of the investigational drug (whichever is shorter); The medication (such as zoledronic acid) for bone metastases related events will not influence on the enrollment;
4. The subjects who previously received major surgery (exclusive of aspiration biopsy) within 8 weeks prior to the initial dosing of the investigational drug, or who are expected to undergo major surgery, or who are in the conditions such as severe unhealed wound, trauma, and ulcer;
5. The subjects who previously received targeted CLDN18.2 therapy (including CLDN18.2 monoclonal antibody, ADC, double antibody, CART);
6. The subjects who have previous serious allergic reactions, or are intolerable to the known component of TST001 or other monoclonal antibodies (including humanized or chimeric antibodies);
7. The subjects who are known to have immediate or delayed hypersensitivity to, be intolerable to or be forbidden from any component of the investigational drugs;
8. The subjects who have previous serious allergic reaction or intolerance to taxane drugs (Cohort D only) or any component of CAPOX (Cohort C and G), PD1 antibody (Cohort G and H) or GP (Cohort F);
9. The subjects in whom symptoms of brain or leptomeningeal metastases are present;

   The subjects with central nerve system (CNS) metastasis who meets the following conditions can be enrolled:

   The subjects with brain metastasis who have not received to any treatment and are asymptomatic, or who are radiologically stable for at least 8 weeks following treatment and do not require hormone or anti epilepsy treatment at least within 8 weeks;
10. The subjects with body cavity effusion (hydrothorax, ascites and pericardial effusion) requiring local treatment or repeated drainage which is not well controlled at the discretion of the investigators;
11. The subjects with concurrent malignant tumors within 3 years other than adequately treated cervical carcinoma in situ, localized squamous cell cancer of the skin, basal cell carcinoma, prostate cancer with no treatment required (with or without resection), ductal carcinoma in situ of the breast, or ≤ T1 urothelial carcinoma (for the dose expansion phase only);
12. Any adverse reactions caused by previous treatment have not resolved to ≤ Grade 1 as per CTCAE v5.0 (exclusive of alopecia and anaemia) before the initial dosing of the investigational drug. If the adverse reaction has no clinical influence, the Sponsor and investigators will decide whether the subject can be enrolled in the study after discussion.
13. The subjects who received growth factor, transfusion or other blood products in treatment of anaemia or decreased platelet within 14 days prior to the initial dose;
14. The subjects who experienced clinically significant cardiovascular and cerebrovascular diseases within 6 months before the initial dosing of the investigational drug, including:

    i. Myocardial infarction, ii. Unstable angina pectoris, iii. Cerebrovascular accident or iv. Other acute uncontrollable cardiovascular diseases; Clinically significant ventricular arrhythmia history (such as ongoing ventricular tachycardia, ventricular fibrillation and torsade de pointes); New York Heart Association (NYHA) Class III or IV congestive cardiac failure; QTc ≥470ms (female) or QTc ≥450ms (male), or medical history or family history of congenital long-QT syndrome (Naring A, 2012); The subjects with heart rhythm disorders requiring the treatment with antiarrhythmic drugs (The subjects who suffer from atrial fibrillation with heart rate controllable more than 1 month before the initial dosing of the investigational drug will be eligible);
15. The subjects who are known to have dihydropyrimidine dehydrogenase (DPD) deficiency. (Note: DPD deficiency screening should be performed according to local requirement.) (The screening will be performed only in the subjects receiving CAPOX.)
16. Subjects with recent gastrointestinal bleeding as evidenced by hematemesis, hematochezia, or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy;
17. The subjects who have evidenced risk of gastric haemorrhage or gastric perforation will be excluded from the study at the discretion of the investigators;
18. The subjects with documented obstruction pyloric and persistent repeated vomiting defined as ≥ 3 episodes within 24 hours;
19. Documented active colitis within 4 weeks prior to study entry, including infectious colitis, radiation colitis and ischemic colitis.
20. History of ulcerative colitis or Crohn's disease;
21. Uncontrolled diarrhea is present;
22. The subjects who are known to have > Grade 1 peripheral sensory neuropathy, unless a lack of deep tendon reflexes is the only neurological abnormality;
23. Active infection requiring systematically intravenous antibiotic therapy within 2 weeks prior to dosing;
24. HIV infection history or positive HIV viral test;
25. The subjects who are known to have the history of hepatitis C or chronic active hepatitis B;

    Except for:
    1. HBV virus carriers or subjects with hepatitis B infection that is stable after medications (HBV-DNA titer should be no more than 1000 copies [cps]/mL or 200 IU/mL); Patients who are not currently on viral suppressive therapy may be eligible and should be discussed with the Medical Monitor and if enrolled, antiviral therapy is required throughout study treatment.
    2. Subjects with hepatitis C infection that is stable after medications (HCV-RNA test negative);
26. Subjects with active autoimmune disorders requiring systemic immunosuppressive therapy within the past 2 years (Subjects with type 1 diabetes mellitus (TD1M), hypothyroidism requiring hormone replacement therapy only, or skin diseases that do not require systemic treatment are eligible);
27. Any disease requiring systemic treatment with corticosteroids (> 10 mg/day prednisone or equivalent drugs) or other immunosuppressive drugs for ≤14 days prior to the first dose of the investigational drug, except for:

    Adrenal replacement steroids (≤10 mg/day prednisone or equivalent drugs) Topical, ophthalmic, intra-articular, intranasal or inhaled corticosteroids with low systemic absorption Preventive corticosteroids (e.g. prevention of contrast media allergy) for short term (≤ 7 days), or corticosteroids for the treatment of non-autoimmune disorders (e.g. delayed type hypersensitivity caused by contactant);
28. Any conditions that the investigators judge that the patient is not appropriate for PD-1 antibody treatment, including but not limited to a history of interstitial lung disease or non-infectious pneumonia, uncontrollable lung diseases, such as pulmonary fibrosis, active pneumonia, etc. (Cohort G and H);
29. Subjects vaccinated live vaccine within 4 weeks before the first dose of the investigational drug;
30. Pregnant or lactating women;
31. Subject with other conditions (such as psychological, geographic or medical conditions) that do not allow them to follow the study schedule and follow-up procedures. Or the subjects who are unsuitable to be enrolled into the study at the discretion of the investigators.

As of protocol version 4.2, enrollment of subjects on the combination protocol no longer requires a positive CLDN18.2 expression result, but enrolled subjects must provide sufficient formalin-fixed paraffin-embedded (FFPE) wax blocks of tumor tissue specimens or at least 10 consecutive white slices) for retrospective CLDN18.2 and PD-L1 testing. (Patients may be enrolled if they have less than 10 specimens, but not less than 7, and meet the requirements of the other inclusion criteria and receive approval from the sponsor's medical ombudsman).

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2020-08-13 (Actual); Primary Completion 2026-06-25 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Participant Safety as characterized by frequency and severity of adverse events(according to NCI CTCAE 5.0). | up to 30 days following last dose.
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Maximum Tolerated Dose (MTD） | up to 28 days following first dose
  The maximum tolerated dose (MTD) is commonly estimated to be the maximum dose that can be determined through DLT of two among 6 subjects administered with TST001 Q2W in 28 days cycles.
Maximum Tolerated Dose (MTD） | up to 21days following first dose
  The maximum tolerated dose (MTD) is commonly estimated to be the maximum dose that can be determined through DLT of two among 6 subjects administered with TST001 once every 3 weeks in 21 days cycles.
Recommended Phase 2 Dose (RP2D) | up to 30 days following last dose
  The RP2D will be determined during the dose expansion stage of the study. RP2D will be determined using available safety and efficacy data.
The incidence and case number of DLT (Dose Limiting Toxicity) in subjects administered with TST001 Q2W in 28 days cycles during observation period | up to 28 days following first dose
  DLT is short for Dose Limiting Toxicity. dose-limiting describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment.
The incidence and case number of DLT (Dose Limiting Toxicity) in subjects administered with TST001 once every 3 weeks in 21 days cycles during observation period | up to 21days following first dose
  DLT is short for Dose Limiting Toxicity. dose-limiting describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment.
Safety and Tolerability of TST001 in combination with other therapies, e.g. CAPOX, paclitaxel, GP, nivolumab as characterized by frequency and severity of adverse events | Up to 30 or 90 days following last dose
  Characterization of TST001 + CAPOX safety profile including frequency and severity of adverse events that are related to treatment.

SECONDARY OUTCOMES:
Area under plasma concentration vs time curve (AUC) for TST001 | up to 30 days following last dose
  Changes in AUC over time in participants with TST001.
Peak plasma concentration (Cmax) for TST001 | up to 30 days following last dose
  Cmax is the maximum plasma concentration.
Time to maximum observed plasma concentration (Tmax) | up to 30 days following last dose
  Tmax is the time in hrs/days it takes to reach Cmax after dosing with TST001
Terminal elimination half life (t1/2) | up to 30 days following last dose
  Time for the plasma level of TST001 to decrease b y 1/2 during the terminal elimination phase.
Immunogenicity | up to 30 days following last dose
  by measurement of Incidence of anti-drug antibodies (ADA)
Objective response rate (ORR) | up to 30 days following last dose
  as measured by RECIST 1.1
Duration of Response (DOR) | up to 30 days following last dose
  DOR is defined as the time from the date of the first response CR (complete remission)/PR (partial remission) (whichever is first recorded) to the date of radiographical progression/death or date of censoring.
Disease Control Rate | up to 30 days following last dose
  DCR: CR+PR+SD
Progression free survival (PFS) and OS | up to 30 days following last dose
  as measured by RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (40):
- China (40):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Guangxi, Guangxi
  - Hainan Provincial People's Hospital, Haikou, Hainan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Heibei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Jinan Central Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Fudan University Shanghai Cance Center, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No